CLINICAL TRIAL: NCT01502462
Title: Prospective Registry of Patients With Isolated Severe Tricuspid Regurgitation
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jong-Min Song, Associate professor, Asan Medical Center
Other Study IDs: Severe_Isol_TR
Record Dates: First submitted 2011-12-29; First posted 2011-12-30 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Tricuspid Regurgitation
Keywords: Clinical course and prognostic factors in patients with severe isolated TR
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Prospective registry for patients with severe isolated tricuspid regurgitation (TR) without significant left-sided valvular or myocardial diseases.

Aim: To evaluate clinical course and prognostic factors of patients with severe isolated TR.

DETAILED DESCRIPTION:
Inclusion criteria Severe isolated TR for more than 6 months

Exclusion criteria

1. Severe mitral and aortic valvular heart disease
2. Age equals to or more than 75 years
3. Malignancy or serious comorbidity with life expectancy < 5years
4. Acute or subacute infective endocarditis requiring antibiotics therapy
5. Untreated hyperthyroidism
6. Constrictive pericarditis
7. Unclosed significant atrial septal defect
8. Previous tricuspid valve surgery
9. Significant coronary artery disease
10. Cardiomyopathy
11. Pregnancy
12. Severe resting pulmonary hypertension(TR Vmax >4.0 m/s)

ELIGIBILITY:
Inclusion criteria

* Severe isolated TR for more than 6 months

Exclusion criteria

1. Severe mitral and aortic valvular heart disease
2. Age equals to or more than 75 years
3. Malignancy or serious comorbidity with life expectancy < 5years
4. Acute or subacute infective endocarditis requiring antibiotics therapy
5. Untreated hyperthyroidism
6. Constrictive pericarditis
7. Unclosed significant atrial septal defect
8. Previous tricuspid valve surgery
9. Significant coronary artery disease
10. Cardiomyopathy
11. Pregnancy
12. Severe resting pulmonary hypertension(TR Vmax >4.0 m/s)

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prospective registry for patients with severe isolated tricuspid regurgitation (TR) without significant left-sided valvular or myocardial diseases.
  Aim: To evaluate clinical course and prognostic factors of patients with severe isolated TR
Sampling Method: Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
all cause death | 5 years

SECONDARY OUTCOMES:
Hospitalization of cardiovascular causes | 5 years
tricuspid valve surgery | 5 years
stroke | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea